CLINICAL TRIAL: NCT06413797
Title: Strengthening Little Cigar and Cigarillo Warnings to Prevent Adolescent Use
Brief Title: Little Cigar and Cigarillo Warnings for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-2455; 5R01CA260822-03 (NIH)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Little Cigars and Cigarillos (LCC) Use
Keywords: cigarette warnings; youth; smoke cigars; nicotine addiction; cancer prevention; Black or African American youth
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FDA warnings + Image (Experimental): Participants will receive FDA-proposed LCC warnings with images
  Interventions: Behavioral: FDA warnings + Image
- FDA Warnings Text-Only Warnings (Experimental): Participants will receive FDA-proposed text-only LCC warnings.
  Interventions: Behavioral: FDA Warnings Text-Only
- Surgeon General Text-Only Warnings (Active Comparator): Participants will receive Surgeon General text-only LCC warnings.
  Interventions: Behavioral: Surgeon General Text-Only Warnings

INTERVENTIONS:
Behavioral: FDA warnings + Image — For six days (days 2-7) participants will be contacted and asked to complete a daily survey. As part of the survey, participants will view FDA-proposed LCC warnings with images at 30% size on a cigarillo package. Participants will be contacted each day to be invited to complete the survey for that day of the study protocol.
  Arms: FDA warnings + Image
Behavioral: FDA Warnings Text-Only — Participants will receive messages including images in 30% size.
  Arms: FDA Warnings Text-Only Warnings
Behavioral: Surgeon General Text-Only Warnings — Participants will receive messages including Surgeon General Text-only Warnings.
  Arms: Surgeon General Text-Only Warnings

SUMMARY:
This study explores the effect of the little cigars and cigarillos (LCC) warnings on youth who currently use, have ever used, or are susceptible to using LCCs. This study will inform the Food and Drug Administration (FDA) implementation of LCC warnings, which can reduce LCC use and lessen tobacco health disparities among youth.

DETAILED DESCRIPTION:
Cigar use exposes youth to the addictive effects of nicotine during a critical developmental period and increases the risk of multiple cancers and premature death. Recent data indicate that cigars are the second most commonly used tobacco product by youth and that past 30-day cigar use is 7.6%, which translates into 1.1 million high school students. Of the three major types of cigars-large cigars, little cigars, and cigarillos-little cigars and cigarillos (LCCs) are the most commonly used in the US, particularly among younger people. LCC use also contributes to tobacco health disparities, as Black or African American youth use cigars more frequently than other youth. In 2016, the Food and Drug Administration (FDA) deemed LCCs subject to FDA regulation, requiring six rotating text-only warning statements to be on LCC packaging. Previous research has examined the effectiveness of LCC warnings in reducing youth willingness to use LCCs.

Research from studies of cigarette warnings suggests that effective LCC warnings should employ images that illustrate negative health effects associated with use and a larger warning label prominently displayed on the pack. Among youth, health warnings on cigarette packs that contain both text statements and images are more effective and engaging than text-only warnings. However, evidence for cigarette warning labels cannot adequately inform implementation of improved LCC warnings for three reasons: 1) there is no evidence on the effectiveness of the FDA-mandated text-only LCC warnings on behavioral intentions or other outcomes among youth 2)courts have ruled that effective tobacco warnings on one type of tobacco product cannot be used to justify warnings on other types of tobacco, and 3) LCC users have different demographic and consumption profiles than cigarette users include more Black/African Americans and use LCCs on fewer days per month.

ELIGIBILITY:
Inclusion Criteria:

1. Members of the recruitment panel (we are partnering with a panel provider for the recruitment of all participants)
2. Agree to provide their honest answers
3. Susceptible to using LCCs, or have ever used little cigars and/or cigarillos, or currently use little cigar and/or cigarillos in the past 30 days
4. Age 15 - 20 years old
5. Currently living in US or US territory
6. Able to complete 2 surveys that take approximately 15 minutes
7. Able to complete a 2-minute survey each day for 6 days
8. Able to verify they are not a bot using CAPTCHA
9. Able to answer a simple, random math question

Exclusion Criteria:

* Not able to verify they are not a bot using Completely Automated Public Turing test to tell Computers and Humans Apart (CAPTCHA).
* Not able to answer a simple, random math question.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 928 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah Ranney, PhD, MA, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowitt SD, Clark SA, Jetsupphasuk M, Jarman KL, Jebai R, Goldstein AO, Cornacchione Ross J, Ranney LM. Examining the influence of descriptors used to market unflavoured cigarillos: an experiment with a sample of youth and young adults from the USA. Tob Control. 2026 Jan 8:tc-2025-059806. doi: 10.1136/tc-2025-059806. Online ahead of print. PMID 41506908
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and screened for study eligibility online between 7/18/2024- 11/25/2024 and invited to in the study once they were determined to be eligible.
Pre-assignment Details: 1,039 potential participants began the baseline survey. Of those, 9 did not consent to participate in the study, and 96 did not complete the baseline questionnaire and were not randomized, and 6 did not meet quality control criteria. 928 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Started | 310 | 309 | 309
Completed | 310 | 309 | 309
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Everyone who enrolled in the study, consented to participate, completed the baseline questionnaire, and was randomized to each condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings | Total
Number analyzed (Participants) | 310 | 309 | 309 | 928
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (1.4) | 18.4 (1.5) | 18.4 (1.5) | 18.5 (1.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 161 | 138 | 143 | 442
  Female | 146 | 170 | 165 | 481
  Unknown | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 68 | 65 | 206
  Not Hispanic or Latino | 236 | 240 | 241 | 717
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 6 | 17
  Asian | 15 | 13 | 17 | 45
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 49 | 52 | 56 | 157
  White | 194 | 192 | 183 | 569
  More than one race | 22 | 12 | 19 | 53
  Unknown or Not Reported | 25 | 32 | 27 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 310 | 309 | 309 | 928

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Use Little Cigars Cigarillos (LCCs)
Description: The average willingness to use score will be measured by the average of the responses to the 2 survey questions scores. Question Scoring is on a scale of 1 to 5, where 1 indicates low willingness to use LCCs, and 5 indicates a willingness to use LCCs score.
Time Frame: Day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 250 | 255 | 236
score on a scale | 2.86 (1.47) | 3.08 (1.39) | 2.99 (1.40)

2. Secondary Outcome: Past 7 Days Little Cigar Use
Description: The number of days in the past 7 days that a participant reported using little cigars, range 0-7. Measured by survey, 1 item.
Time Frame: Day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 250 | 256 | 236
number of days | 1.92 (2.62) | 1.86 (2.60) | 1.88 (2.59)

3. Secondary Outcome: Past 7 Days Cigarillo Use
Description: The number of days in the past 7 days that a participant reported using cigarillos, range 0-7. Measured by survey, 1 item.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 249 | 256 | 236
number of days | 1.93 (2.57) | 1.86 (2.41) | 1.82 (2.33)

4. Secondary Outcome: Little Cigar and Cigarillos (LCCs) Susceptibility
Description: The average susceptibility to little cigar and cigarillo (LCC) use measured with the average of 3 survey item scores. Question scoring is on a scale of 1 to 4, where 1 indicates high susceptibility and 4 indicates low susceptibility to LCCs.
Time Frame: Day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 250 | 256 | 236
score on a scale | 2.33 (0.97) | 2.49 (0.91) | 2.46 (0.95)

5. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: The cognitive elaboration score is measured by survey with 1 item. Question scoring is on a scale of 1 to 6, where 1 indicates that the participant has low cognitive elaboration about the health risks of LCCs and 6 indicates that a participant has high cognitive elaboration about smoking LCCs.
Time Frame: Day 2
Population: Participants who responded to the scale at the time point of interest, day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 218 | 229 | 205
units on a scale | 3.78 (1.60) | 3.90 (1.64) | 3.91 (1.60)

6. Secondary Outcome: Warning Negative Affect/Worry
Description: Warning negative affect/worry is measured by survey with 1 item. Question scoring is on a scale of 1 to 5, where 1 indicates low worry due to the warning and 5 indicates high worry due to the warning.
Time Frame: Day 2
Population: Participants who responded to the scale at the time point of interest, day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 218 | 229 | 205
units on a scale | 3.79 (1.16) | 3.85 (1.23) | 3.61 (1.26)

7. Secondary Outcome: Knowledge of Little Cigar and Cigarillo (LCC) Harms
Description: Knowledge of LCC harms will be measured by 12 items the survey. Scores can range from 0 to 12 and indicate the number of questions out of 12 about LCC harms that participants answered correctly.
Time Frame: Day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 250 | 256 | 236
score on a scale | 10.06 (2.63) | 10.12 (2.46) | 9.71 (2.82)

8. Secondary Outcome: Beliefs About Little Cigar and Cigarillo (LCC) Harms
Description: The average score on beliefs about LCC harms measured with 10 items by survey, are an average of the responses to the 10 questions. Belief scoring is on a scale of 1 to 5, where 1 indicates strong disagreement with statements about the health harms of LCCs and 5 indicates strong agreement with the statements about the health harms of LCCs.
Time Frame: Day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 249 | 256 | 236
score on a scale | 4.30 (0.58) | 4.31 (0.54) | 4.24 (0.59)

9. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 3
Population: Participants who responded to the scale at the time point of interest, day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 231 | 240 | 227
units on a scale | 3.97 (1.46) | 4.08 (1.50) | 3.74 (1.64)

10. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 4
Population: Participants who responded to the scale at the time point of interest, day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 238 | 233 | 216
units on a scale | 3.88 (1.59) | 3.94 (1.52) | 3.74 (1.65)

11. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 5
Population: Participants who responded to the scale at the time point of interest, day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 225 | 238 | 217
units on a scale | 4.00 (1.53) | 4.08 (1.54) | 3.88 (1.64)

12. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 6
Population: Participants who responded to the scale at the time point of interest, day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 230 | 222 | 217
units on a scale | 4.01 (1.58) | 4.05 (1.59) | 3.78 (1.67)

13. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 7
Population: Participants who responded to the scale at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 218 | 208 | 209
units on a scale | 3.98 (1.54) | 4.11 (1.50) | 3.83 (1.70)

14. Secondary Outcome: Cognitive Elaboration About Risk of Little Cigar and Cigarillo Use
Description: as for outcome 5
Time Frame: Day 8
Population: Participants who responded to the scale at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 250 | 256 | 236
units on a scale | 4.12 (1.55) | 3.99 (1.52) | 4.00 (1.60)

15. Secondary Outcome: Warning Negative Affect/Worry
Description: as for outcome 6
Time Frame: Day 3
Population: Participants who responded to the scale at the time point of interest, day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 231 | 240 | 227
units on a scale | 4.02 (1.04) | 3.42 (1.24) | 3.48 (1.26)

16. Secondary Outcome: Warning Negative Affect/Worry
Description: as for outcome 6
Time Frame: Day 4
Population: Participants who responded to the scale at the time point of interest, day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 238 | 233 | 216
units on a scale | 4.03 (1.15) | 3.55 (1.25) | 3.65 (1.20)

17. Secondary Outcome: Warning Negative Affect/Worry
Description: as for outcome 6
Time Frame: Day 5
Population: Participants who responded to the scale at the time point of interest, day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 225 | 238 | 217
units on a scale | 4.00 (1.13) | 3.52 (1.38) | 3.36 (1.29)

18. Secondary Outcome: Warning Negative Affect/Worry
Description: as for outcome 6
Time Frame: Day 6
Population: Participants who responded to the scale at the time point of interest, day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 230 | 222 | 217
units on a scale | 4.02 (1.08) | 3.72 (1.23) | 3.71 (1.23)

19. Secondary Outcome: Warning Negative Affect/Worry
Description: as for outcome 6
Time Frame: Day 7
Population: Participants who responded to the scale at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
Number analyzed (Participants) | 218 | 208 | 209
units on a scale | 3.90 (1.13) | 3.79 (1.15) | 3.79 (1.16)

ADVERSE EVENTS:
Time Frame: Low risk study, no adverse event data collected
Description: Low risk study, no adverse event data collected
Arm/Group | FDA Warnings + Image | FDA Warnings Text-Only Warnings | Surgeon General Text-Only Warnings
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT06413797/Prot_SAP_000.pdf